CLINICAL TRIAL: NCT05395611
Title: Exhaled Breath Particles as Biomarkers for Diagnosing, Prognosticating and Evaluating of Non Small Cell Lung Cancer
Brief Title: Exhaled Breath Particles in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PExCaP
Record Dates: First submitted 2022-05-10; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer; Lung Adenocarcinoma; Squamous Cell Lung Cancer
Keywords: Exhaled Breath Particles; PExA; Lung cancer; Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled breath particles (EBP) Blood samples Tumor tissue and surrounding non tumor lung tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer: Patients with primary non small cell lung cancer listed for tumor resection. EBP, plasma and lung tumor tissue will be collected for protein profiling.
  Collection of EBP will be done at 2 time points before and after surgery. Collection of plasma will be done at 2 time points before and after surgery. Collection of lung/tumor tissue will be done at the time of surgery
  Interventions: Other: EBPcollected using the PExA device.
- Control: Patients without lung cancer matched according to age and smoking history (control cohort) Collection of EBP will be done at one time point. Collection of plasma will be done at one time point.
  Interventions: Other: EBPcollected using the PExA device.

INTERVENTIONS:
Other: EBPcollected using the PExA device. — The PExA device is a non invasive device that collect particles in exhaled air

SUMMARY:
Lung cancer (CaP) is the leading cause of cancer related deaths on a global level. Early diagnosis is vital for survival and life quality of the affected patients, yet lung cancer is often diagnosed at advanced stages, causing poor five-year survival rates. Exhaled breath particles (EBP) and particle flow rate (PFR) collected by the particles in exhaled air (PExA) system is a safe and easily reproducible non-invasive method for gaining insight into the molecular environment of the distal airways. EBP and PFR have been found useful in detection of other airway diseases such as acute respiratory distress syndrome (ARDS), primary graft dysfunction (PGD) and bronchiolitis obliterans syndrome (BOS). It has been shown that particles found in EBP reflect the general composition of respiratory tract lining fluid (RTLF) and that biomarkers found in EBP correlate to proteins that can be found in both bronchoalveolar lavage fluid (BALF) and plasma. Particle flow rate (PFR) has been found to differ between patients with lung cancer compared to control patients. In the present study the investigators aim to collect EBP samples and measure PFR from patients with primary lung cancer and from control patients. EBPs are collected for molecular analysis. The investigators aim to identify biomarkers for diagnosing, predicting prognosis of and evaluating surgical treatment of non small cell lung cancer.

DETAILED DESCRIPTION:
EBP samples and measurements of PFR will be collected from patients with primary non-small cell lung cancer (NSCLC) at Skåne University Hospital (SUS) Lund. Measurements will be done at 2 time points, before and after surgical resection for NSCLC.

EBP samples will be collected at one time point from a matched (by age and smoking history) control cohort.

Blood samples will be collected from both cohorts, at the same time points as the EBP/PFR measurements.

Tumor tissue and healthy adjacent lung tissue will be collected from lung cancer patients with tumors greater than 3 cm in diameter on preoperative computed tomography.

The purpose of this clinical trial is to identify non-invasive means of diagnosing NSCLC at earlier stages. The PExA method is not associated with any risks and has potential minimize hospitalization associated with more invasive methods that are in clinical practice today, such as bronchoscopy and biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung cancer with clinical Tumor, Node, Metastasis (TNM) up to cT3N1M0 according to TNM 7th edition
* Able to take instructions and perform the standardized breathing maneuver

Exclusion Criteria:

* Dementia
* Severe neurological disease
* Drug abuse
* Heart failure New York Heart Association (NYHA) Classification, NYHA class III or IV
* Ejection fraction < 50 %
* S-creatinine > 140 µmol/L
* Poorly regulated diabetes mellitus

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with primary lung cancer and listed for tumor resection. Patients without lung cancer.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Protein concentration in exhaled breath particles (EBP) | Before surgery for NSCLC
  EBPs are collected on membranes and analyzed in regards to protein concentration and abundance
Protein concentration in exhaled breath particles (EBP) | After surgery for NSCLC (2 weeks - 36 months)
  EBPs are collected on membranes and analyzed in regards to protein concentration and abundance
Protein concentration in exhaled breath particles (EBP) | In patients without NSCLC (control cohort). (0- 2 weeks)
  EBPs are collected on membranes and analyzed in regards to protein concentration and abundance

SECONDARY OUTCOMES:
Particle flow rate (PFR) expressed as particles/liter of exhaled air | Before surgery for NSCLC
  Particle flow rate (PFR) has recently been shown to differ significantly between patients suffering from respiratory diseases such as bronchiolitis obliterans syndrome (BOS) and covid-19 compared to healthy controls. PFR will be measured from patients with primary lung cancer and control patients to investigate if PFR can be used to distinguish between the two groups and thus help diagnosing lung cancer in earlier stages.
Particle flow rate (PFR) expressed as particles/liter of exhaled air | After surgery for NSCLC (2 weeks - 36 months)
  Particle flow rate (PFR) has recently been shown to differ significantly between patients suffering from respiratory diseases such as bronchiolitis obliterans syndrome (BOS) and covid-19 compared to healthy controls. PFR will be measured from patients with primary lung cancer and control patients to investigate if PFR can be used to distinguish between the two groups and thus help diagnosing lung cancer in earlier stages.
Particle flow rate (PFR) expressed as particles/liter of exhaled air | In patients without NSCLC (control cohort). (0- 2 weeks)
  Particle flow rate (PFR) has recently been shown to differ significantly between patients suffering from respiratory diseases such as bronchiolitis obliterans syndrome (BOS) and covid-19 compared to healthy controls. PFR will be measured from patients with primary lung cancer and control patients to investigate if PFR can be used to distinguish between the two groups and thus help diagnosing lung cancer in earlier stages.
Protein expression in plasma | Before surgery for NSCLC
  Concentration and composition of proteins will be measured in plasma from lung cancer patients
Protein expression in plasma | After surgery for NSCLC (2 weeks - 36 months)
  Concentration and composition of proteins will be measured in plasma from lung cancer patients
Protein expression in plasma | In patients without NSCLC (control cohort). (0- 2 weeks)
  Concentration and composition of proteins will be measured in plasma from healthy control patients
Protein expression in tissue | During surgery for NSCLC. (0- 2 weeks)
  Concentration and composition of proteins will be measured in tumor tissue and the surrounding lung tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt, MD, PhD, Principal Investigator — Region Skåne, Lund University
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenlo M, Hyllen S, Silva IAN, Bolukbas DA, Pierre L, Hallgren O, Wagner DE, Lindstedt S. Increased particle flow rate from airways precedes clinical signs of ARDS in a porcine model of LPS-induced acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2020 Mar 1;318(3):L510-L517. doi: 10.1152/ajplung.00524.2019. Epub 2020 Jan 29. PMID 31994907
- [Background] Broberg E, Hyllen S, Algotsson L, Wagner DE, Lindstedt S. Particle Flow Profiles From the Airways Measured by PExA Differ in Lung Transplant Recipients Who Develop Primary Graft Dysfunction. Exp Clin Transplant. 2019 Dec;17(6):803-812. doi: 10.6002/ect.2019.0187. Epub 2019 Oct 11. PMID 31615381
- [Background] Behndig AF, Mirgorodskaya E, Blomberg A, Olin AC. Surfactant Protein A in particles in exhaled air (PExA), bronchial lavage and bronchial wash - a methodological comparison. Respir Res. 2019 Sep 26;20(1):214. doi: 10.1186/s12931-019-1172-1. PMID 31558154
- [Background] Broberg E, Andreasson J, Fakhro M, Olin AC, Wagner D, Hyllen S, Lindstedt S. Mechanically ventilated patients exhibit decreased particle flow in exhaled breath as compared to normal breathing patients. ERJ Open Res. 2020 Feb 10;6(1):00198-2019. doi: 10.1183/23120541.00198-2019. eCollection 2020 Jan. PMID 32055633